CLINICAL TRIAL: NCT07265167
Title: An Open-label, Randomized, Fasting, Single-dose, Oral Administration, 2- Sequence, 2-period, Crossover Study to Evaluate Bioequivalence Study Between YHP2406 and YHR2501 in Healthy Subjects
Brief Title: Bioequivalence Study Between YHP2406 and YHR2501 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yuhan Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: YHP2406-102
Record Dates: First submitted 2025-11-23; First posted 2025-12-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Healthy Subjects
Keywords: Pharmacokinetics; Bioequivalence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A(RT) (Experimental): 31 subjects, Cross-over, Single dose YHR2501 on period 1, Single dose of YHP2406 on period 2
  Interventions: Drug: YHP2406; Drug: YHR2501
- B(TR) (Experimental): 31 subjects, Cross-over, Single dose of YHP2406 on period 1, Single dose of YHR2501 on period 2
  Interventions: Drug: YHP2406; Drug: YHR2501

INTERVENTIONS:
Drug: YHP2406 — Test drug: YHP2406, Comparator: YHR2501
Drug: YHR2501 — Test drug: YHP2406, Comparator: YHR2501

SUMMARY:
A randomized, open-label, single-dose, 2-sequence, 2-period, crossover clinical trial to investigate the bioequivalence between YHP2406 and YHR2501 in healthy volunteers

DETAILED DESCRIPTION:
62 healthy subjects will be randomized to one of the 2 groups in the same ratio.

Subjects in group 1 will be administered "comparator" and "YHP2406" by crossover design on period 1, 2. Subjects in group 2 will be administered "YHP2406" and "comparator" by crossover design on period 1, 2.

ELIGIBILITY:
Inclusion Criteria:

* BMI 18-30 kg/m2
* Those without clinically significant congenital or chronic diseases

Exclusion Criteria:

* Those who have participated in a bioequivalence study or other clinical trials and have been administered with investigational products in 6 months prior to the first administration.
* Others who are judged ineligible to participate in the trial by the principal investigator.
* Female volunteers who are pregnant, suspected to be pregnant or breastfeeding.

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2025-10-18 (Actual); Primary Completion 2025-10-20 (Actual); Study Completion 2025-11-04 (Actual)

PRIMARY OUTCOMES:
Area under the plasma drug concentration-time curve [AUCt] | 0-8 hours
  Area under the plasma drug concentration-time curve [AUCt] of Amoxicillin & Clavulanic acid
Maximum plasma concentration [Cmax] | 0-8 hours
  Maximum plasma concentration [Cmax] of Amoxicillin & Clavulanic acid

SECONDARY OUTCOMES:
Area under the plasma drug concentration-time curve from time 0 to infinity [AUCinf] | 0-8 Hours
  Area under the plasma drug concentration-time curve from time 0 to infinity [AUCinf] of Amoxicillin & Clavulanic acid
Area under the plasma drug concentration-time curve/Area under the plasma drug concentration-time curve from time 0 to infinity [AUCt/AUCinf] | 0-8 Hours
  Area under the plasma drug concentration-time curve/Area under the plasma drug concentration-time curve from time 0 to infinity [AUCt/AUCinf] of Amoxicillin & Clavulanic acid
Time of peak concentration [Tmax] | 0-8 Hours
  Time of peak concentration [Tmax] of Amoxicillin & Clavulanic acid
Terminal phase of half-life [t1/2] | 0-8 Hours
  Terminal phase of half-life [t1/2] of Amoxicillin & Clavulanic acid

CONTACTS AND LOCATIONS:
Overall Officials: Seoung Hyun Kang, Principal Investigator — H Plus Yangji Hospital
Locations (1):
- H Plus Yangji Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No